CLINICAL TRIAL: NCT03605992
Title: Compliance, Viability and Effectiveness of Home Based Cardiac Rehabilitation: a Randomised Trial
Brief Title: Home-based Cardiac Rehabilitation: Compliance and Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Raquel Rodrigues Britto, Full Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMMinasGerais
Record Dates: First submitted 2018-03-21; First posted 2018-07-30 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Cardiac Disease
Keywords: Rehabilitation; Coronary artery disease; Home-based; Randomized Controlled Trial; Protocol
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Rehabilitation (Experimental): Home-based cardiac rehabilitation that includes the components of education and physical exercises mainly unsupervised and oriented by telephone.
  Interventions: Other: Home-based Rehab
- CentreRehabilitation (Active Comparator): Traditional cardiac rehabilitation offered at the outpatient centre including components of education and physical exercises mainly supervised.
  Interventions: Other: CentreRehab

INTERVENTIONS:
Other: Home-based Rehab — This intervention will have the duration of 12 weeks, with a total of 60 sessions: 2 supervised and 58 at home (to complete five exercise's sessions for week).
  Arms: Home-based Rehabilitation
Other: CentreRehab — This intervention will last 12 weeks, with a total of 60 sessions: 24 supervised and 36 at home (to complete five exercise's sessions for week).
  Arms: CentreRehabilitation

SUMMARY:
The proposal of this study is to verify if it is feasible and effective to offer a home based cardiac rehabilitation program, that includes the components of health education and physical exercises mostly unsupervised and oriented by telephone and to compare the treatment adherence, the effects in the functional capacity, and the control of coronary risk factors in relation to the traditional cardiac rehabilitation offered mostly supervised and center based.

DETAILED DESCRIPTION:
This study will be developed with patients with coronary disease submitted to angioplasty or myocardial revascularization surgery, provided they are considered of low and moderate risk for the practice of physical exercise of moderate intensity, according to the risk stratification proposed by the American Association of Cardiovascular and Pulmonary Rehabilitation. Volunteers will be recruited at the outpatient at the University Hospital's Cardiac Rehabilitation Centre. The study will be made in conformity with the CONSORT guidelines for non-pharmacological interventions. After being invited to the study, the volunteer whose accept the participation and sign the consent form will be randomized into two different groups: Traditional cardiac rehabilitation (mostly supervised) and Telerehabilitation (mostly unsupervised). The randomization will be made through the www.randomization.com website in blocks of four volunteers each. A blind researcher will evaluate participants before and after test, and will fulfill the database.

Intervention The parameters for the exercise prescription will be the same for both groups. Exercise sessions will be constituted of 5-10 minutes of warm up, 40 minutes of aerobic activity with heart rate between 60 and 80% of the heart rate reserve, and 5-10 minutes of cool down. The educational sessions will be given to both groups in six meetings with 40 minutes each, and items regarding the control of risk factors and treatment of cardiovascular diseases will be approached. After the period of 12 weeks of intervention all participants will be stimulated to continue to practice physical exercises at home or at the community, and they will be invited to a re-evaluation after three months.

Groups:

Traditional cardiac rehabilitation as control group (CentreRehab) The CentreRehab group will be made supervised exercises and health educational activities, personally at cardiac rehabilitation centre. This intervention will last 12 weeks, with a total of 60 sessions: 24 supervised and 36 at home (to complete five exercise's sessions for week). The participants of this group will be oriented to fulfill a training diary with information regarding the frequency of the exercises, the presence of symptoms, and the use of the scale of perceived exertion during exercises at home.

Home-based cardiac rehabilitation (HomeRehab) The participants of the HomeRehab group will make the exercise mostly at home. There will be weekly phone calls, in person educational sessions, and monthly meetings to check the execution of the previous stage, solve doubts, or identify the presence of symptoms or undesirable effects. This intervention will have the duration of 12 weeks, with a total of 60 sessions: 2 supervised and 58 at home (to complete five exercise's sessions for week).

In the first week, all individuals of HomeRehab group will receive a training regarding the use of the monitoring equipment. A heart rate monitor with the heart rate zone individually calculated will be given to the participant at the first session of the face-to-face training to monitoring exercises at home. Furthermore, all participants of this group will use a step counter (pedometer) to stimulate the execution of the exercises as well as training diary to be fulfilled with information regarding the frequency of the exercises, the presence of symptoms during the exercise, the perceived exertion, and the number of daily steps. The monthly meetings will take place to the educational activity, and to verify if the exercises and fulfilment of the training diary are correct as well as to clarify any kind of the participant's doubts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary disease submitted to angioplasty or myocardial revascularization surgery, or that had a heart attack, provided they are considered of a low and moderate risk for the practice of physical exercise of moderate intensity according to the stratification for the risk of events during a cardiovascular rehabilitation program
2. Clinical stability, according with the medical evaluation;
3. Residents of the Belo Horizonte's metropolitan region.

Exclusion Criteria:

1. Recent cardiac event or clinical decompensation (<1month);
2. Presence of peripheral arterial occlusive disease with limitation degree that prevents the test of maximum exercise (emergence of claudication before the maximum cardiorespiratory fatigue);
3. Presence of chronic pulmonary disease (i.e. Chronic Obstructive Pulmonary Disease, pulmonary fibrosis, and pulmonary arterial hypertension of pre capillary etiology);
4. History of ventricular fibrillation or sustained ventricular tachycardia in the last year;
5. Presence of high risk criteria during the ergometric test;
6. Physical, cognitive, or social limitation that prevent the participation in a physical exercise program, and the comprehension of the use of the monitoring device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in adherence on CR sessions | after 3 and 6 months of the intervention
  it will be analyzed by the percentage of participants which completed the minimum of 75% of the sessions

SECONDARY OUTCOMES:
Cost | after 3 and 6 months of the intervention
  total sum of the costs of each procedure applied to different groups considering the table of payments for procedures and services of the hospital.
Usability | For TeleRehab group after 3 months of the intervention
  it will be analyzed using the System Usability Scale (SUS) after 3 months. The System Usability Scale (SUS) is a widely used self-administered instrument for the evaluation of usability of a wide range of products and user interfaces. The main value of the SUS is that it provides a single reference score for the participants' view of the usability of a product or service.
  The SUS's scores vary in a value between zero and 100. A SUS's scores higher than 68 is considered above average, and any value below.
Change in morbidity | after 3 and 6 months of the intervention
  It will be evaluated through a survey to identify the number of hospitalizations, complications, and presence of clinical events during the period of 3 and 6 months.
Change in quality of life | At baseline, after 3 and 6 months
  Quality of life will be assessed by the Short-Form 36 (SF-36) questionnaire, a generic questionnaire, easy to administrate, that considers the individual perception about its own health status. It's composed by 36 items, divides in eight domains: physical functioning, physical role functioning, bodily pain, general health perceptions, vitality, social role functioning, emotional role functioning, and mental health. Data will be analyzed from the transformation of the answers in each domain in a scale from zero (0) to one hundred (100). This questionnaire won't have a cut point, and the analysis is made based in the hit score, resulting in a worse or better general health state.
Change in scores of depression | At baseline, after 3 and 6 months
  The Patient Health Questionnaire-9 (PHQ-9) is a simple test, used for depression screening. The PHQ-9 is an instrument that has nine items, disposed in a scale of four points, from zero (not once) to three (almost every day), with a score that varies from zero to 27, to asses frequency of signs and symptoms of depression in the last two weeks. It is estimated, as a positive indicator of major depression, a value equal or higher than 10.
Change in functional capacity | At baseline, after 3 and 6 months
  Functional Capacity will be analyzed using the Incremental Shuttle walk test, a walk test that evaluates functional capacity through the analysis of the walked distance at incremental shuttle walk test in meters.
Change in level of physical activity | At baseline, after 3 and 6 months
  Score at the Duke Activity Status Index, a questionnaire developed to evaluate functional capacity mostly in patients with cardiovascular diseases. This questionnaire is composed of 12 items, which asses daily life activities such as personal hygiene, locomotion, domestic tasks, sexual function, and recreation, with the respective metabolic costs. Each item has a specific weight, based on its metabolic cots. The weight of the positive answers is summed up in order to obtain a total score that goes from zero to 58.2. The higher the punctuation, higher the functional capacity.
Change in Blood pressure | At baseline, after 3 and 6 months
  Systolic and diastolic blood pressure measured at rest
Change in Waist circumference | At baseline, after 3 and 6 months
  measurement of the waist circumference in centimeters.
Change in fasting blood glucose | At baseline, after 3 and 6 months
  assessed through blood exams, as mg/dL
Change in glycated hemoglobin | At baseline, after 3 and 6 months
  values, in %, will be assessed through blood tests.
Change in total cholesterol | At baseline, after 3 and 6 months
  In mg/dL, will be assessed through blood tests.
Change in knowledge about coronary artery disease | At baseline, after 3 and 6 months
  Will be analyzed using the CADE-Q SV. This questionnaire was designed to be a true/false/I don't know questionnaire, with 20 items (4 in each domain). Each correct answer equals to 1 point; therefore, the maximum score possible is 20 overall, 4 by domain, and 1 per item.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel R Britto, Post doc, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mezzani A, Hamm LF, Jones AM, McBride PE, Moholdt T, Stone JA, Urhausen A, Williams MA; European Association for Cardiovascular Prevention and Rehabilitation; American Association of Cardiovascular and Pulmonary Rehabilitation; Canadian Association of Cardiac Rehabilitation. Aerobic exercise intensity assessment and prescription in cardiac rehabilitation: a joint position statement of the European Association for Cardiovascular Prevention and Rehabilitation, the American Association of Cardiovascular and Pulmonary Rehabilitation, and the Canadian Association of Cardiac Rehabilitation. J Cardiopulm Rehabil Prev. 2012 Nov-Dec;32(6):327-50. doi: 10.1097/HCR.0b013e3182757050. PMID 23103476
- [Result] Varnfield M, Karunanithi M, Lee CK, Honeyman E, Arnold D, Ding H, Smith C, Walters DL. Smartphone-based home care model improved use of cardiac rehabilitation in postmyocardial infarction patients: results from a randomised controlled trial. Heart. 2014 Nov;100(22):1770-9. doi: 10.1136/heartjnl-2014-305783. Epub 2014 Jun 27. PMID 24973083
- [Result] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Result] Coutinho-Myrrha MA, Dias RC, Fernandes AA, Araujo CG, Hlatky MA, Pereira DG, Britto RR. Duke Activity Status Index for cardiovascular diseases: validation of the Portuguese translation. Arq Bras Cardiol. 2014 Apr;102(4):383-90. doi: 10.5935/abc.20140031. Epub 2014 Feb 17. PMID 24652056
- [Result] Santos IS, Tavares BF, Munhoz TN, Almeida LS, Silva NT, Tams BD, Patella AM, Matijasevich A. [Sensitivity and specificity of the Patient Health Questionnaire-9 (PHQ-9) among adults from the general population]. Cad Saude Publica. 2013 Aug;29(8):1533-43. doi: 10.1590/0102-311x00144612. Portuguese. PMID 24005919
- [Result] Ghisi GLM, Sandison N, Oh P. Development, pilot testing and psychometric validation of a short version of the coronary artery disease education questionnaire: The CADE-Q SV. Patient Educ Couns. 2016 Mar;99(3):443-447. doi: 10.1016/j.pec.2015.11.002. Epub 2015 Nov 7. PMID 26610390
- [Derived] Lima AP, Nascimento IO, Oliveira ACA, Martins THS, Pereira DAG, Britto RR. Home-Based Cardiac Rehabilitation in Brazil's Public Health Care: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Nov 7;8(11):e13901. doi: 10.2196/13901. PMID 31697246
- See also: American Association for Cardiovascular and Pulmonary Rehabilitation. Guidelines for Cardiac Rehabilitation and Secondary Prevention Programs. 5th ed. Champaign.Human Kinetics Publishers; 2013. — http://www.humankinetics.com/products/all-products/guidelines-for-cardiac-rehabilitation-and-secondary-prevention-programs-5th-edition-with-web-resource
- See also: CICONELLI, R.M. et al. Brazilian Portuguese version of the SF-36. A reliable and valid quality of life outcome measure. Rev. Bras. Reumatol., v.39, n.3, p.143-50, 1999. — https://toneurologiaufpr.files.wordpress.com/2013/03/questionc3a1rio-de-qualidade-de-vida-sf36-traduc3a7c3a3o-e-validac3a7c3a3o.pdf